CLINICAL TRIAL: NCT03255408
Title: Role of Cerebral Blood Flow on Ventilatory Stability During Sleep in Normoxia and Intermittent Hypoxia
Brief Title: Cerebral Blood Flow and Ventilatory Responses During Sleep in Normoxia and Intermittent Hypoxia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Marc Poulin, PhD, DPhil, Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: REB13-0880
Record Dates: First submitted 2017-08-06; First posted 2017-08-21 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Obstructive Sleep Apnea of Adult; Hypoxia, Brain; Sleep Apnea; Sleep Disorder; Stroke; Blood Pressure; Endothelial Dysfunction; Oxidative Stress
MeSH Terms: conditions — Hypoxia, Brain; Sleep Apnea Syndromes; Sleep Wake Disorders; Stroke | interventions — Core Binding Factors; Cerebrovascular Circulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CBF Lowering and Normoxia Sleep (Active Comparator): Study participants will take drug lowering Cerebral Blood Flow (CBF) and sleep under room air i.e. normoxia exposure.
  Interventions: Drug: Drug Lowering Cerebral Blood Flow (CBF) and Normoxia Sleep
- CBF Lowering and IH Sleep (Experimental): Study participants will take drug lowering Cerebral Blood Flow (CBF) and sleep under Intermittent Hypoxia (IH) exposure.
  Interventions: Drug: Drug Lowering CBF and Intermittent Hypoxia Sleep
- Placebo and Normoxia Sleep (Sham Comparator): Study participants will take Placebo that has no effect on Cerebral Blood Flow (CBF) and sleep under room air i.e. normoxia exposure.
  Interventions: Drug: Placebo and Normoxia Sleep
- Placebo and IH Sleep (Placebo Comparator): Study participants will take Placebo that has no effect on Cerebral Blood Flow (CBF) and sleep under Intermittent Hypoxia (IH) exposure.
  Interventions: Drug: Placebo and Intermittent Hypoxia Sleep

INTERVENTIONS:
Drug: Drug Lowering Cerebral Blood Flow (CBF) and Normoxia Sleep — The study participants will take Cerebral Blood Flow (CBF) lowering drug and sleep under Normoxia Exposure
  Other Names: Cerebral Blood Flow changes and Normoxia Sleep
  Arms: CBF Lowering and Normoxia Sleep
Drug: Drug Lowering CBF and Intermittent Hypoxia Sleep — The study participants will take Cerebral Blood Flow (CBF) lowering drug and sleep under Intermittent Hypoxia (IH) Exposure
  Other Names: CBF changes and Intermittent Hypoxia Sleep
  Arms: CBF Lowering and IH Sleep
Drug: Placebo and Normoxia Sleep — The study participants will take Placebo and sleep under Normoxia Exposure
  Other Names: Cerebral Blood Flow (CBF) with Placebo in Normoxia Sleep
  Arms: Placebo and Normoxia Sleep
Drug: Placebo and Intermittent Hypoxia Sleep — The study participants will take Placebo and sleep under Intermittent Hypoxia (IH) Exposure
  Other Names: CBF with Placebo in Intermittent Hypoxia Sleep
  Arms: Placebo and IH Sleep

SUMMARY:
A prospective double blind, placebo-controlled, randomized cross-over trial to evaluate the effect of lowering cerebral blood flow on the ventilatory chemoreflexes (acute hypoxic and hypercapnic ventilatory responses).

DETAILED DESCRIPTION:
The investigators will explore the relationship between changes in Cerebral Blood Flow (CBF) and ventilatory chemoreflexes i.e. Acute Ventilatory Response to Hypoxia (AHVR) and Acute Hypercapnic Ventilatory Response (HCVR) before, during and after sleep under normoxic conditions and sleep accompanied by isocapnic Intermittent Hypoxia (IH) among healthy human study participants.

A pharmacological intervention will be utilized to manipulate the CBF in a randomized order. The study participants will also be randomly assigned the order to sleep either under normoxia or IH exposure. The experiments will be separated from one another with an interval of sufficient drug and IH exposure washout period. The venous blood samples and urinary samples will be collected for the vascular biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* 18 - 45 years of age
* Living in Calgary for the past one year
* Have no medical condition or should not be taking any blood pressure medications.
* The participant should not be lactose intolerant

Exclusion Criteria:

* Cerebrovascular, cardio-respiratory, renal and metabolic diseases
* Bleeding disorders and upper gastrointestinal diseases e.g. peptic ulcer disease
* Pregnancy, obese and sleep-disordered breathing
* Drug allergies to non-steroidal anti-inflammatories
* Currently smoking

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in cerebral blood flow and ventilatory chemoreflexes | ~18 months (from the starting time of recruiting study participants)
  The relationship between changes in cerebral blood flow (CBF) and ventilatory chemoreflexes (acute hypoxic and hypercapnic ventilatory responses) before and after sleeping under normoxia and intermittent hypoxia exposure among healthy human study participants.
Cerebral blood flow responses and ventilatory chemoreflexes during sleep | ~18 months (from the starting time of recruiting study participants)
  The relationship between cerebral blood flow (CBF) changes and ventilatory chemoreflexes (acute hypoxic and hypercapnic ventilatory responses) during sleep under normoxia and intermittent hypoxia exposure among healthy human study participants.

SECONDARY OUTCOMES:
Changes in reactive oxygen species and vascular biomarkers | ~24 months (from the starting time of recruiting study participants)
  The changes in vascular biomarkers such as nitric oxide, reactive oxygen species and exosome analysis or urinary prostaglandins before and after sleep under normoxia and intermittent hypoxia exposure with cerebral blood flow changes.